CLINICAL TRIAL: NCT01025011
Title: Non- Invasive Measurement of the Absolute Hemoglobin Value in the Retinal Arteries of Anemic and Healthy Subjects Using a New Approach
Brief Title: Non-invasive Measurement of Hemoglobin in Retinal Arteries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Triemli Hospital (Other)
Responsible Party: Prof Yves Robert, Stadtpital Triemli (Triemli Hospital)
Other Study IDs: D20028132
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-11

CONDITIONS: Healthy Subjects; Anemia
Keywords: retinal hemoglobin concentration; non-invasive hemoglobin measurement
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy volunteers, anemic patients: healthy volunteers from the eye and gynecology department pregnant patients with anemia
  Interventions: Device: Fundus photography, cubital blood draw

INTERVENTIONS:
Device: Fundus photography, cubital blood draw — blood draw from a cubital vein to measure hemoglobin concentration taking a fundus photography with a Nidek AFC-230, no pupil dilation needed

SUMMARY:
The purpose of this study is to test a new non-invasive tool to measure hemoglobin in retinal arteries.

DETAILED DESCRIPTION:
To our knowledge no tool exists that allows for direct collection of hemoglobin data in the eye. In many eye diseases (especially diabetic and hypertensive retinopathy as well as in retinal vessel occlusions) retinal circulation is modified. Knowing hemoglobin concentration on the site of the pathology will give us further information about the pathogenesis of this diseases and may provide a new possibility in therapy.

The purpose of this study is to test a new non-invasive tool to measure hemoglobin in retinal arteries. Healthy volunteers from the eye clinic and pregnant otherwise healthy patients of the gynecological department of the Triemli Hospital, Zurich, as well as anemic gynecological patients that show up for a check-up are included.

Hemoglobin will be quantified by a blood draw of a cubital vein. Using a Fundus Camera (Nidek AFC-230) pictures of the fundus will be taken from each study patient. Afterwards the study investigator selects a retinal artery of interest which will be used for measuring the hemoglobin concentration. Intensity of the green channel of the camera chip is determined with the aid of the law of Lambert-Beer.

Absolute Hemoglobin concentration is calculated in relation to the vessel volume.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* pregnant patients from the Triemli Hospital that came for a routine check up
* anemic patients of the same dept with various gynecological tumors

Exclusion Criteria:

* any known retinal eye disease
* poor fundus picture quality due to fixtion problems or too small pupil or media intransparency
* not willing to participate in a study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects from the eye clinic of Triemli Hospital anemic and pregnant patients from the gynecology department, Triemli Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Correlation of hemoglobin concentration measured in a cubital vein and in a non invasive way using hemoglobinometry in the retinal veins | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yves Robert, Prof MD, Principal Investigator — Triemli Hospital
Locations (1):
- Stadtpital Zürich, Triemli Hospital, Zurich, Canton of Zurich, Switzerland